CLINICAL TRIAL: NCT07243886
Title: Mobile-based Obstetric Monitoring for Pregnancies Complicated by Hypertension and/or Diabetes (MOM-HD): a Type II Hybrid Implementation-Effectiveness Trial
Brief Title: Mobile-based Obstetric Monitoring for Pregnancies Complicated by Hypertension and/or Diabetes (MOM-HD)
Acronym: MOM-HD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Dhulikhel Hospital (Other); Institute for Implementation Science and Health (Unknown)
Responsible Party: Principal Investigator, Shristi Rawal, PhD, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro2025001611
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Gestational Diabetes; Hypertensive Disorder of Pregnancy
Keywords: pregnancy; telemonitoring; mHealth; GDM; HDP; Nepal; implementation
MeSH Terms: conditions — Diabetes, Gestational; Toxemia | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: In total, 864 participants (432 patients with HDP and 432 patients with GDM will be randomly assigned in a 1:1 fashion to one of two treatment conditions: either (i) MOM-HD program+ standard care or (ii) standard care only from enrolment into pregnancy till six weeks postpartum. Random permuted blocks of sizes 4 or 6 will be employed using statistical software to prevent treatment imbalance and ensure that participants are allocated to each group equally.
Masking Description: The allocation sequence will be concealed from the research nurse and participants using sequentially numbered opaque sealed envelopes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MOM-HD Intervention Group (Experimental): In addition to standard care, participants in the intervention group will use the MOM-HD telemonitoring program, which includes patient education, a blood pressure (BP) monitor and/or glucometer, and a mobile app for uploading daily BP/blood glucose (BG) readings. Women with GDM will receive both devices; those with HDP will receive a BP monitor. The MOM-HD app transfers readings via Bluetooth, provides reminders for BP/BG testing, and allows providers to review data through a secure portal. Nurses will conduct biweekly tele-visits to review results, address concerns, and connect patients with OB/GYNs or dieticians as needed. The goal is to improve self-monitoring, patient-provider communication, and timely clinical decision-making, ultimately enhancing maternal and neonatal outcomes. Both groups continue standard antenatal care, with MOM-HD designed to evaluate the added benefit of telemonitoring.
  Interventions: Behavioral: MOM-HD
- Standard Care Group (Active Comparator): In standard care, pregnant women with HDP and GDM are required to attend hospitals more frequently than the usual antenatal schedule, typically adding 6-8 extra visits for closer monitoring. The maternal-fetal medicine specialist customizes the follow-up schedule, often requiring visits every two weeks until 35 weeks, then weekly. During these visits, patients undergo tests such as ultrasounds, urine dipsticks for proteinuria, and BP/BG monitoring, with results recorded in paper booklets assigned to each patient. Additionally, women are encouraged to regularly monitor their BP and/or BG (fasting and 2-hour post-prandial) at home or at the nearest health post. GDM patients also consult a dietitian and physical therapist to develop a personalized diet and exercise plan based on pre-pregnancy weight and disease severity. OB/GYN physicians monitor BP/BG levels and adjust medications accordingly. Follow-up BP/BG testing is conducted six weeks postpartum.
  Interventions: Other: Standard Care

INTERVENTIONS:
Behavioral: MOM-HD — Participants will receive education and training on proper BP and/or BG monitoring and will be provided a BP monitor and/or glucometer with strips. They will be asked to use the MOM-HD mobile app to measure and record daily BP (until 6 weeks postpartum) and, for women with GDM, fasting and 2-hour postprandial BG (until delivery). Readings are automatically uploaded via Bluetooth to a provider portal and reviewed daily by a nurse. Participants will receive automated reminders, instant feedback on readings, and educational materials via the app. They will participate in biweekly tele-visits with a nurse to review readings, discuss symptoms, and receive counseling on lifestyle, diet, and care plans.
  Arms: MOM-HD Intervention Group
Other: Standard Care — Pregnant women with HDP and GDM will receive standard antenatal care, which includes more frequent hospital visits (6-8 extra), ultrasound, urine dipstick, BP/BG monitoring with paper record booklets, dietary and physical activity counseling, and OB/GYN follow-up. GDM patients will consult with a dietitian and physical therapist. Postpartum follow-up includes BP/BG testing at 6 weeks.
  Arms: Standard Care Group

SUMMARY:
Hypertensive disorders during pregnancy (HDP) and gestational diabetes (GDM) are among the leading complications in pregnancy, significantly contributing to global maternal and fetal morbidity and mortality. (1,2,3) Effective management of HDP and GDM hinges on regular monitoring of blood pressure (BP) and blood glucose (BG) to ensure adequate control and timely interventions for maternal and fetal well-being. Telemonitoring offers a promising and cost-effective alternative by enabling pregnant individuals to monitor BP and BG at home and share real-time results with healthcare providers, facilitating informed clinical decision-making and timely interventions.

Here the investigators propose to conduct a Hybrid Type II Effectiveness-Implementation Randomized Controlled Trial (RCT) to assess the effectiveness and evaluate the implementation of the MOM-HD (Mobile-based Obstetric Monitoring for Hypertension and/or Diabetes) program, a mobile app-based perinatal telemonitoring program, in real-world clinical settings in Nepal. To address the study aims, the investigators will recruit 864 women who are newly diagnosed with HDP and GDM from three metropolitan hospitals and randomly assign them to either (i) MOM-HD + standard care or (ii) standard care alone, from enrolment in pregnancy to 6 weeks postpartum. Primary and secondary clinical outcomes will be assessed at delivery, and at 6 weeks postpartum. The investigators hypothesize that compared to standard care, the use of MOM-HD in addition to standard care will result in lower systolic BP levels, lower incidence rate for the composite adverse perinatal outcome of either perinatal loss, neonatal intensive care unit admission, primary cesarean delivery or labor induction, and lower proportion of days with elevated systolic BP or BG readings between recruitment and 6 weeks postpartum. A convergent mixed-methods approach will be used to assess implementation and maintenance outcomes using the RE-AIM framework (4), and economic sustainability will be assessed by collecting primary cost data.

DETAILED DESCRIPTION:
This is a Mobile-based Obstetric Monitoring for Hypertension and/or Diabetes (MOM-HD)2 program, which includes a patient-facing mobile app for uploading BP/BG data, a provider-facing web portal for viewing patient data, and biweekly tele-visits with a study nurse.

This study aims to utilize an implementation science framework to implement and comprehensively evaluate a mobile app-based perinatal telemonitoring program within real-world clinical settings. Collaborating with government and hospital stakeholders, the investigators will employ a theory-informed multi-faceted implementation strategies: (a) Train patients and family members, and provide continuous technical support (via mobile app) for at-home BP and/or BG monitoring; (b) Provide financial assistance for at-home BP and/or BG monitoring; (c) Technical assistance, audit, and feedback to the providers; and (d) Institutionalizing and sustaining the program through advisory boards at each hospital.

Study Objective and Aims

Primary Goal:

To conduct a hybrid type II effectiveness-implementation randomized controlled trial (RCT) to evaluate the impact of MOM-HD on clinical outcomes and assess its implementation in real-world settings in Nepal.

Specific aims:

* Aim 1: Assess the effectiveness of MOM-HD + standard care compared to standard care alone via a multi-center randomized controlled trial.
* Aim 2: Assess implementation outcomes of the MOM-HD using the RE-AIM framework at the patient, provider, and health system levels.
* Aim 3: Conduct a comprehensive costing analysis and economic evaluation of the MOM-HD.

Study Design

This is a type II hybrid effectiveness-implementation study conducted as a multi-site randomized controlled trial in three metropolitan hospitals in Nepal: 1) Paropakar Maternity and Women's Hospital (PMWH), 2) Dhulikhel Hospital in Dhulikhel, and 3)Nobel Medical College & Teaching Hospital in Biratnagar.

The MOM-HD telemonitoring program will consist of patient education/ training, provision of a BP monitor and/or glucometer and strips, a mobile app where BP/BG data can be uploaded, a provider-facing web portal for monitoring patient data, as well as biweekly tele-visits with a study nurse. Participants with HDP and/or GDM in the intervention group will be enrolled in the MOM-HD program from enrollment to 6 weeks postpartum.

Overall, this study aims to evaluate the effectiveness and implementation of the MOM-HD intervention, while providing insights into the costs associated with implementing the intervention in a real-world setting.

Study Duration

The study is expected to last up to 5 years. Participants will be followed from 24-30 weeks' gestation until 6 weeks postpartum.

Sample Size

A total of 864 participants (432 with HDP and 432 with GDM).

Randomization

Participants will be randomized in a 1:1 ratio to either the intervention group (MOM-HD plus standard care) or the control group (standard care alone).

Study Population: See section Eligibility

Measurements

* Primary and Secondary Outcomes: See section Outcome Measures
* Implementation Outcomes: Using the RE-AIM framework (4), the study will assess Reach (e.g., proportion and characteristics of participants engaged), Adoption (provider uptake), Implementation (fidelity, facilitators, barriers), and Maintenance (sustainability and costs).

Intervention: See section Arms and Interventions

Research Method: Mixed-method and Randomized Clinical Trial

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women receiving antenatal care at RCT site
* Diagnosed with one of the following: Chronic hypertension (sustained systolic BP ≥140 mm Hg and/or diastolic BP ≥90 mm Hg, or on antihypertensive treatment before 20 weeks of gestation) or Gestational hypertension (sustained systolic BP ≥140 mm Hg and/or diastolic BP ≥90 mm Hg after 20 weeks of gestation)
* Gestational diabetes
* Age 18 years or older
* Access to a smartphone

Exclusion Criteria:

* Multifetal pregnancies
* Apparent communication difficulties (e.g., hearing, speech, or cognitive impairments), as judged by research assistants
* Unable to understand the Nepali language
* Requires hospital admission due to severe illness
* Declines to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 864 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2030-02-28 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean systolic BP from recruitment to delivery (continuous) | Post-treatment (at delivery)
  Mean systolic BP levels will be calculated based on data abstracted from the MOM-HD app (home measurements) and medical records (hospital measurements).
Mean systolic BP averaged over 6 weeks postpartum | Post-treatment (6 weeks postpartum)
  Mean systolic BP levels will be calculated based on data abstracted from the MOM-HD app (home measurements) and medical records (hospital measurements). Values averaged from discharge to 6 weeks postpartum.
Rate of composite adverse perinatal outcome (categorical; either perinatal loss, neonatal intensive care unit admission, primary cesarean delivery or labor induction) | Post-treatment (at delivery)
  Perinatal loss, neonatal intensive care unit admission, primary cesarean delivery or labor induction will be abstracted from medical records.
Proportion of days with elevated blood pressure (BP) or blood glucose (BG) readings (above clinical target ranges) between recruitment and delivery (continuous) | Post-treatment (at delivery)
  BP levels or BG levels will be abstracted from the MOM-HD app (home measurements) and medical records (hospital measurements), and proportion of days with elevated readings (out of total number of days with valid measurements) will be calculated.
Proportion of days with elevated blood pressure (BP) or blood glucose (BG) readings (above clinical target ranges) over 6 weeks postpartum (continuous) | Post-treatment (at delivery)
  BP levels or BG levels will be abstracted from the MOM-HD app (home measurements) and medical records (hospital measurements), and proportion of days with elevated readings (out of total number of days with valid measurements) will be calculated, spanning from discharge to 6 weeks postpartum

SECONDARY OUTCOMES:
Mean diastolic BP from recruitment to delivery (continuous) | Post-treatment (at delivery)
  Mean diastolic BP levels will be calculated based on data abstracted from the MOM-HD app (home measurements) and medical records (hospital measurements).
Mean diastolic BP over the 6 weeks postpartum (continuous) | Post-treatment (6 weeks postpartum)
  Mean diastolic BP levels will be calculated based on data abstracted from the MOM-HD app (home measurements) and medical records (hospital measurements).
Mean fasting BG levels from recruitment to delivery (continuous; only among women with GDM) | Post-treatment (at delivery)
  Mean BG levels will be calculated based on data abstracted from the MOM-HD app (home measurements) and medical records (hospital measurements).
Mean postprandial BG levels from recruitment to delivery (continuous; only among women with GDM) | Post-treatment (at delivery)
  Mean BG levels will be calculated based on data abstracted from the MOM-HD app (home measurements) and medical records (hospital measurements).
Perinatal loss (present/ absent) | Post-treatment (at delivery)
  Perinatal loss (present/ absent) will be abstracted from medical records
Neonatal intensive care unit admission (present/absent) | Post-treatment (at delivery)
  Neonatal intensive care unit admission (present/ absent) will be abstracted from medical records.
Primary cesarean delivery (present/absent) | Post-treatment (at delivery)
  Primary cesarean delivery (present/absent) will be abstracted from medical records.
Induction of labor (present/ absent) | Post-treatment (at delivery)
  Induction of labor (present/absent) will be abstracted from medical records.
Need for medication ( present/ absent) | Post-treatment (at delivery)
  Medication initiation will be abstracted from medical records
Pre-term birth ( present/ absent) | Post-treatment (at delivery)
  Gestational age at delivery will be abstracted from medical records
Hospital admissions ( present/ absent) | Post-treatment (at delivery)
  Hospital admissions will be abstracted from medical records

OTHER OUTCOMES:
App usage (Intervention group only) | at six weeks postpartum
  The MOM-HD app will keep a usage record for each of the individual app feature(s) used (e.g., BP/BG), time of day the app/feature was used, and time spent in each feature.
App compliance ( Intervention group only) | at six weeks postpartum
  Self-monitoring frequency data, such as the number of BP/BG entries in the app over the entire monitoring period, will be recorded for each participant in the intervention group. This is the actual number of app entries divided by the expected app entries multiplied by 100).
Usability ( Intervention group only) | at six weeks postpartum
  The System Usability Scale, (5) a 10-item 5-point Likert scale questionnaire will be administered to assess the perceived usability of the MOM-HD app.

CONTACTS AND LOCATIONS:
Overall Officials: Shristi Rawal, PhD, Principal Investigator — Rutgers School of Health Professions

IPD SHARING:
Plan to Share IPD: Yes
After information that could identify the participant has been removed, de-identified information collected for this research may be shared and made publicly available as required by the National Institute of Health (NIH). The investigators will include the clinical data of those participants who provide consent for sharing their data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Release of data will occur approximately 12 months following the end of the study. Study data will be available to the research community without end date.
Access Criteria: The investigator will only share or make publicly available de-identified data collected for this research. The investigators will include the clinical data of those participants who provide consent for sharing their data.

REFERENCES:
- [Background] Say L, Chou D, Gemmill A, Tuncalp O, Moller AB, Daniels J, Gulmezoglu AM, Temmerman M, Alkema L. Global causes of maternal death: a WHO systematic analysis. Lancet Glob Health. 2014 Jun;2(6):e323-33. doi: 10.1016/S2214-109X(14)70227-X. Epub 2014 May 5. PMID 25103301
- [Background] Murray SR, Reynolds RM. Short- and long-term outcomes of gestational diabetes and its treatment on fetal development. Prenat Diagn. 2020 Aug;40(9):1085-1091. doi: 10.1002/pd.5768. Epub 2020 Jul 1. PMID 32946125
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547